CLINICAL TRIAL: NCT06854354
Title: Intervention for Human Papillomavirus Vaccine Acceptance in Mexican Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Univeristario Benemerita Universidad Autonoma de Puebla (Other)
Collaborators: Benemerita Universidad Autónoma de Puebla (Unknown); Facultad de Enfermería (Unknown)
Responsible Party: Principal Investigator, Gabriela Iveth Martínez Figueroa, Master in Nursing, Hospital Univeristario Benemerita Universidad Autonoma de Puebla
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SIEP/ME/111/2021
Record Dates: First submitted 2025-02-22; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Papillomavirus Infections; Papillomavirus Vaccines
Keywords: papillomavirus infections; human papillomavirus vaccine; Intervention for mothers; behavioral change
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial (RCT), which was divided into an Experimental Group (EG) and a Control Group (CG), where the independent variable was the intervention "Vaccine for HPV prevention", which contained the knowledge of HPV and the vaccine, interpersonal influences, benefits and perceived barriers of the HPV vaccine, likewise, the dependent variable was the acceptance of the HPV vaccine. The intervention was a single-blind approach, with a test-retest model, measuring the variables before and after the educational intervention.
Who Masked: Participant
Masking Description: Participants were unaware of the group to which they belonged and the interventions to the other group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The intervention was designed using the theory-based approach to designing interventions, using MPS middle-range theory. This approach focused on managing HPV vaccine acceptance in mothers of girls aged 9 to 12 years. The intervention was structured in five steps: understanding the problem, identifying aspects susceptible to change, establishing intervention strategies, selecting modes and doses of administration, and developing a procedures manual. In addition, the results of a qualitative study were integrated to identify mothers' needs for information about the vaccine. The intervention focused on increasing knowledge and acceptance of the vaccine, decreasing perceived barriers. It was validated through the Content Validity Coefficient (CVC), obtaining values that indicated high validity. It was delivered through a private Facebook group, where educational materials were provided and participants completed questionnaires to assess their level of knowledge. The intervention consiste
  Interventions: Behavioral: HPV Prevention Vaccine
- Control Group (Placebo Comparator): The CG did not have an educational intervention, nor the use of any placebo, the test instruments were applied and a month after this, they were invited to a virtual platform where they were asked to answer again the measurement instruments, once obtained the filling of the questionnaires they were invited and provided the user guide that allowed them to participate and learn about the Facebook group, as well as view the educational materials, to obtain the same benefits as the GE
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: HPV Prevention Vaccine — The educational intervention was implemented through a private Facebook group, facilitating access to HPV vaccine information. A user guide was provided and profiles were verified for authenticity using a non-duplicity algorithm. Prior to access, mothers completed questionnaires to assess their knowledge, beliefs and acceptance. The intervention lasted four weeks and included four modules with videos, handouts and infographics. The first session provided information on HPV, its transmission and prevention. The second highlighted the benefits of the vaccine and debunked myths. The third showed testimonials from mothers who had their daughters vaccinated. The last session was a videoconference with group dynamics to resolve doubts. The sessions were held weekly and access and duration were monitored within the group. After finishing, the group was temporarily closed to avoid biases in the second measurement, allowing free access to the contents.
  Arms: Experimental Group
Other: Placebo — The CG did not have an educational intervention, nor the use of any placebo, the test instruments were applied and a month after this, they were invited to a virtual platform where they were asked to answer again the measurement instruments, once obtained the filling of the questionnaires they were invited and provided the user guide that allowed them to participate and learn about the Facebook group, as well as view the educational materials, to obtain the same benefits as the GE
  Arms: Control Group

SUMMARY:
Randomized clinical trial with two groups, with a test-retest model, with single-blind approach, using a probabilistic sampling and the population was mothers of girls aged 9 to 12 years from a public elementary school in the state of Puebla. The objective was to determine the effect of the intervention "Vaccine for HPV Prevention" aimed at the acceptance of the HPV vaccine in mothers of girls aged 9 to 12 years old in the urban area of the State of Puebla.

DETAILED DESCRIPTION:
Introduction: Human papillomavirus is a serious health problem worldwide, being immunization the viable prevention strategy to combat the infection, however, there is a low acceptance of the vaccine in mothers to immunize their daughters, derived from social, economic, cultural and educational aspects. Objective: To determine the effect of the intervention "Vaccine for HPV Prevention" aimed at the acceptance of the HPV vaccine in mothers of girls aged 9 to 12 years old in the urban area of the State of Puebla. Methodology: Randomized clinical trial with two groups, with a test-retest model, with a single-blind approach, a probabilistic sampling was used and the population was 10 mothers of girls from 9 to 12 years old from a public elementary school in the state of Puebla.

ELIGIBILITY:
Inclusion Criteria:

* Women from 20 to 59 years old.
* Mothers of girls from 9 to 11 years old.
* Who agree to participate in the study.
* Who know how to read and write.
* Who have an electronic device (cell phone, tablet or computer).
* That they have access to social networks such as WhatsApp and Facebook.
* That they have an internet connection.

Exclusion Criteria:

* Mothers with a history of CACU and/or HPV infection in themselves or a family member.
* Mothers who have received information about CACU, HPV and/or the HPV vaccine at least one month prior to the educational intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
knowledge of HPV | 3 months
  To measure knowledge of the HPV vaccine, the valid and reliable questionnaire designed by Xolocotzi, Marín, Gómez & Valenzuela (2011), applied in the Mexican context, was used. For the purposes of this study only dimension four called prevention, diagnosis and treatment was used, consisting of 8 items (28, 29, 30, 31, 33, 33, 33, 34 and 35), with a dichotomous response pattern of true and false. The result translates into, the greater the number of correct answers, the greater the knowledge of the HPV vaccine, the reliability of the instrument was through the Kuder-Richardson 20 coefficient, obtaining an rtt = .833.
Positive and negative beliefs about HPV and the vaccine | 3 months
  A valid and reliable instrument, adapted to the Mexican context, was used to measure the factors that influence the acceptance or refusal of the HPV vaccine in mothers of girls. It consists of 40 questions grouped into six dimensions: general information about HPV (items 9-15, Cronbach's alpha .60); beliefs about HPV and the vaccine (items 16-31, alpha .58); information mechanisms (items 1-8, alpha .80); perceived benefits (items 20-22, alpha .74); barriers (items 23-26, 39-40, alpha .74); and acceptance of the vaccine (items 32-38, alpha .90). Responses are presented on a dichotomous scale (Yes/No) or in a four-point Likert format (1=strongly disagree, 4=strongly agree). The results are standardized on a 100-point scale, where higher values reflect greater knowledge, perceived benefits or acceptance of the vaccine. Overall, the instrument has a Cronbach's Alpha of .70, indicating acceptable internal reliability.
Acceptance of the human papillomavirus vaccine | 3 months
  A valid and reliable instrument, adapted to the Mexican context, was used to measure the factors that influence the acceptance or refusal of the HPV vaccine in mothers of girls. It consists of 40 questions grouped into six dimensions: general information about HPV (items 9-15, Cronbach's alpha .60); beliefs about HPV and the vaccine (items 16-31, alpha .58); information mechanisms (items 1-8, alpha .80); perceived benefits (items 20-22, alpha .74); barriers (items 23-26, 39-40, alpha .74); and acceptance of the vaccine (items 32-38, alpha .90). Responses are presented on a dichotomous scale (Yes/No) or in a four-point Likert format (1=strongly disagree, 4=strongly agree). The results are standardized on a 100-point scale, where higher values reflect greater knowledge, perceived benefits or acceptance of the vaccine. Overall, the instrument has a Cronbach's Alpha of .70, indicating acceptable internal reliability.

SECONDARY OUTCOMES:
Acceptability of human papillomavirus vaccine | 12 months
  Mothers should increase their intention to vaccinate their daughters against the human papillomavirus (HPV) with the bivalent or quadrivalent vaccine by approaching their nearest health centers. The impact of this intervention will be measured through vaccination application rates, calculated based on attendance lists from the educational institutions involved. The vaccination rate will be determined by dividing the number of vaccinated students by the total number of eligible students listed in these institutions.

CONTACTS AND LOCATIONS:
Overall Officials: Vianet Nava Navarro, PhD, Study Director — School of Nursing - Benemerita Universidad Autónoma de Puebla
Locations (1):
- Faculty of Nursing - Benemerita Universidad Autonoma de Puebla, Puebla City, Puebla, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
the intervention is still undergoing replication to test its effectiveness and efficacy, so the principal investigators continue to modify doses and modes of delivery.

REFERENCES:
- [Background] Susanto T, Rif'ah EN, Susumaningrum LA, Rahmawati I, Yunanto RA, Evayanti NLP, Utami PAS. Human papillomavirus vaccine acceptability among healthcare workers, parents, and adolescent pupils: a pilot study in public health centers of Bali, Indonesia. Germs. 2020 Sep 1;10(4):184-194. doi: 10.18683/germs.2020.1204. eCollection 2020 Sep. PMID 33134196
- [Background] Ryan C, Duvall KL, Weyant EC, Johnson KR, Wood D. Human Papillomavirus Vaccine Uptake, Knowledge, and Acceptance for Youth: A Systematic Review of Appalachia. J Community Health. 2018 Jun;43(3):616-624. doi: 10.1007/s10900-018-0500-6. PMID 29564684
- [Background] Rabiu KA, Alausa TG, Akinlusi FM, Davies NO, Shittu KA, Akinola OI. Parental acceptance of human papillomavirus vaccination for adolescent girls in Lagos, Nigeria. J Family Med Prim Care. 2020 Jun 30;9(6):2950-2957. doi: 10.4103/jfmpc.jfmpc_102_20. eCollection 2020 Jun. PMID 32984154
- [Background] Joseph NP, Bernstein J, Pelton S, Belizaire M, Goff G, Horanieh N, Freund KM. Brief Client-Centered Motivational and Behavioral Intervention to Promote HPV Vaccination in a Hard-to-Reach Population: A Pilot Randomized Controlled Trial. Clin Pediatr (Phila). 2016 Aug;55(9):851-9. doi: 10.1177/0009922815616244. Epub 2016 Mar 10. PMID 26968631
- [Background] Odunyemi FT, Ndikom CM, Oluwatosin OA. Effect of Nursing Intervention on Mothers' Knowledge of Cervical Cancer and Acceptance of Human Papillomavirus Vaccination for their Adolescent Daughters in Abuja - Nigeria. Asia Pac J Oncol Nurs. 2018 Apr-Jun;5(2):223-230. doi: 10.4103/apjon.apjon_75_17. PMID 29607384
- [Background] Grandahl M, Paek SC, Grisurapong S, Sherer P, Tyden T, Lundberg P. Parents' knowledge, beliefs, and acceptance of the HPV vaccination in relation to their socio-demographics and religious beliefs: A cross-sectional study in Thailand. PLoS One. 2018 Feb 15;13(2):e0193054. doi: 10.1371/journal.pone.0193054. eCollection 2018. PMID 29447271
- [Background] Galbraith-Gyan KV, Lechuga J, Jenerette CM, Palmer MH, Moore AD, Hamilton JB. HPV vaccine acceptance among African-American mothers and their daughters: an inquiry grounded in culture. Ethn Health. 2019 Apr;24(3):323-340. doi: 10.1080/13557858.2017.1332758. Epub 2017 May 29. PMID 28553758
- [Background] Degarege A, Krupp K, Srinivas V, Ibrahimou B, Marlow LAV, Arun A, Madhivanan P. Determinants of attitudes and beliefs toward human papillomavirus infection, cervical cancer and human papillomavirus vaccine among parents of adolescent girls in Mysore, India. J Obstet Gynaecol Res. 2018 Nov;44(11):2091-2100. doi: 10.1111/jog.13765. Epub 2018 Aug 16. PMID 30117218
- [Background] Cory L, Cha B, Ellenberg S, Bogner HR, Hwang WT, Smith JS, Haggerty A, Morgan M, Burger R, Chu C, Ko EM. Effects of Educational Interventions on Human Papillomavirus Vaccine Acceptability: A Randomized Controlled Trial. Obstet Gynecol. 2019 Aug;134(2):376-384. doi: 10.1097/AOG.0000000000003379. PMID 31306313
- [Background] Cheruvu VK, Bhatta MP, Drinkard LN. Factors associated with parental reasons for "no-intent" to vaccinate female adolescents with human papillomavirus vaccine: National Immunization Survey - Teen 2008-2012. BMC Pediatr. 2017 Feb 13;17(1):52. doi: 10.1186/s12887-017-0804-1. PMID 28193249
- [Background] Allen JD, Hollander J, Gualtieri L, Alarcon Falconi TM, Savir S, Agenor M. Feasibility of a twitter campaign to promote HPV vaccine uptake among racially/ethnically diverse young adult women living in public housing. BMC Public Health. 2020 Jun 1;20(1):830. doi: 10.1186/s12889-020-08824-0. PMID 32487045